CLINICAL TRIAL: NCT05086913
Title: A Comparison of Self-help Lifestyle Modification Delivered by a Smartphone App and Booklets in Managing Depressive Symptoms: a Pilot Randomised Controlled Trial.
Brief Title: Self-help Lifestyle Medicine App and Booklets for Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY017
Record Dates: First submitted 2021-10-09; First posted 2021-10-21 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Depression
Keywords: Depression; Self-help; Lifestyle Medicine; Well-being
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle medicine smartphone app (Experimental): The app group will receive an app to facilitate lifestyle modification such as video demonstrations of physical activity, diet recommendations, stress and sleep management.
  Interventions: Other: Lifestyle medicine smartphone app
- lifestyle medicine booklets (Experimental): The booklet group will receive 8 lifestyle medicine and psychoeducation booklets with identical content with the lifestyle medicine app.
  Interventions: Other: Lifestyle medicine smartphone booklets
- waitlist control (Sham Comparator): The waitlist control group will receive access to the lifestyle medicine app and booklets at the end of the study.
  Interventions: Other: Waitlist control

INTERVENTIONS:
Other: Lifestyle medicine smartphone booklets — Participants will receive a pocket size 6-page booklet weekly over 8 weeks that covers 8 lifestyle medicine, mental health and CBT themes including stress, relaxation, diet, exercise, sleep hygiene, worry management, mindfulness, and positive psychology, and guides participants to set and meet short term and long-term goals.
  Arms: lifestyle medicine booklets
Other: Lifestyle medicine smartphone app — The lifestyle medicine app offers 8 modules with identical content as the wellness booklets, in addition to videos, relaxation, exercise and cooking demonstrations, daily challenges, record of goals, and ecological momentary assessments of diet, physical activity, sleep, stress and mood.
  Arms: Lifestyle medicine smartphone app
Other: Waitlist control — The waitlist control group will receive access to the lifestyle medicine app and booklets at the end of the study.
  Arms: waitlist control

SUMMARY:
This study aims to compare self-help lifestyle medicine (LM) delivered by a smartphone app and booklets in managing depressive symptoms in a Chinese population.

This study is a randomised controlled trial. First, informed consent will be obtained from potential participants. Around 90 eligible participants will be randomly assigned to either the LM app group, the LM booklet group, and the waitlist control group, in a ratio of 1:1:1. The app group will receive an app to facilitate lifestyle modification such as video demonstrations of physical activity, diet recommendations, stress and sleep management. The booklet group will receive 8 LM booklets with identical content with the LM app. The waitlist control group will receive access to the app and booklets at the end of the study. The whole intervention lasts 8 weeks. Participants will also receive 2 messages per week from the researcher to check and prompt motivation and adherence. Participants will complete assessment before, immediately after intervention, at one month and 12-week follow up.

DETAILED DESCRIPTION:
As lifestyle plays an important role in the pathogenesis of depression, lifestyle medicine (LM) emerges as a new way to alleviate depressive symptoms (Sarris & O'Neil, 2016). Booklets have been shown as an inexpensive and effective delivery modality of lifestyle modification among individuals with physical conditions (Wong, Chair & Wong, 2017). Meanwhile, a recent meta-analysis supports the efficacy of mobile applications in improving depressive symptoms (Linardon, Cujipers, Carlbring, Messer & Fuller-Tyszkiewicz, 2019). Notably, the efficacy of lifestyle intervention using booklets and app have not been compared. This pilot study can inform the field about the efficacy of lifestyle intervention using two self-help delivery modalities and offer new ways to better managing depressive symptoms.

This study will be a randomised controlled trial comparing self-help LM delivered by a smartphone app and booklets in improving depression. For a pilot study, a sample size of 12 per group is recommended (Julious, 2005). Considering an estimation of 20% attrition at the three assessment time points, the final sample size is 90, with 30 participants in each group.

The LM booklet group will receive a pocket size 6-page booklet weekly that covers 8 lifestyle medicine themes including stress, relaxation, diet, exercise, sleep hygiene, worry management, mindfulness, and positive psychology. Exercises based on cognitive behavioural therapy and guidance to set and meet short term and long-term goals are featured in the booklets. The booklet series is reviewed by a panel of experts including clinical psychologists, psychiatrists, dietitians, physical trainers, and traditional Chinese Medicine practitioners. The app group will receive access to a mobile app that offers 8 modules with identical content as the wellness booklets, in addition to videos, relaxation, exercise and cooking demonstrations, daily challenges and record of goals. The waitlist control group will receive access to the app and booklets at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with elevated depressive symptoms as defined by PHQ-9 score 10 or above
* Hong Kong residents
* Aged 18 or above
* Able to read Chinese and type in Chinese or English
* Have an Internet-enabled mobile device (iOS or Android operating system)

Exclusion Criteria:

* Pregnancy;
* Using medication or psychotherapy for depression;
* Currently participating in other psychological intervention studies;
* Cognitive impairment;
* Having unsafe conditions and are not recommended for physical activity or a change in diet by physicians;
* Self-disclosure of any major psychiatric, medical, or neurocognitive disorders that make participation unsuitable or may interfere with the adherence of the lifestyle modification;
* Any suicidal ideation (scoring above 2 in item 9 in BDI-II) Participants with any urgent health necessity were excluded and referred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | baseline, immediately post-intervention, 4-week and 12-week follow-up
  The PHQ-9, a 20-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Self-developed survey | Baseline
  A self-developed survey will collect information including demographic information (e.g., age, gender, level of education, working industry, relationship status, and location of residence), substance use, body mass index (BMI), rest-activity pattern, and social rhythms, etc.
Change in the World Health Organization 5-item Well-Being Index | baseline, immediately post-intervention, 4-week and 12-week follow-up
  This is a 5-item measure of global subjective well-being. The internal consistency prior to treatment was 0.86.
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | baseline, immediately post-intervention, 4-week and 12-week follow-up
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the Perceived Stress Scale (PSS) | baseline, immediately post-intervention, 4-week and 12-week follow-up
  The PSS measures the perceived amount of stress experienced over the past month.
Change in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) | baseline, immediately post-intervention, 4-week and 12-week follow-up
  The GAD-7, a 7-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of anxiety over the past two weeks on a 4-point scale, "0" (not at all) to "4" (nearly every day).
Change in the Sheehan Disability Scale (SDS) | baseline, immediately post-intervention, 4-week and 12-week follow-up
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in the Health-Promoting Lifestyle Profile (HPLP II) | baseline, immediately post-intervention, 4-week and 12-week follow-up
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
Change in the International Physical Activities Questionnaire - Chinese version (IPAQ-C) | baseline, immediately post-intervention, 4-week and 12-week follow-up
  Participants' sitting time, walking time and moderate and vigorous physical activity are assessed by 5 questions from the short form of the International Physical Activity Questionnaire - Chinese version. Participants' engagement in brief strength and stamina-enhancing activity were assessed by asking the number of days they engaged in physical activity while seated and standing in the last seven days.
Change in the Insomnia Severity Index (ISI) | baseline, immediately post-intervention, 4-week and 12-week follow-up
  The ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong